CLINICAL TRIAL: NCT01471678
Title: An Open-label, Randomized, Single Dose, Four-Period Crossover Study to Compare the Bioavailability of Fixed Dose Combination Capsule Formulations of Dutasteride and Tamsulosin Hydrochloride (0.5 mg/0.2 mg) With 10% and 15% of Enteric Coated Pellets With Harnal-D Tablets and Harnal Capsules Co-administered With Dutasteride (0.5 mg) Soft Gel Capsules in Healthy Male Subjects of North East Asian Ancestry
Brief Title: Bioavailability of Two Combination Products of Dutasteride (0.5mg) and Tamsulosin Hydrochloride (0.2mg) in Asian Males.
Acronym: ARI115707
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 115707
Record Dates: First submitted 2011-10-13; First posted 2011-11-16 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Prostatic Hyperplasia
Keywords: Cross-over design; Pilot bioequivalence; North east Asian ancestry; GI198745; Tamsulosin hydrochloride; healthy male subjects; Bioequivalence; Dutasteride
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Dutasteride; Tamsulosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fixed dose combination product (Experimental): Fixed Dose Combination capsule containing dutasteride 0.5mg and tamsulosin 0.2 mg
  Interventions: Drug: Dutasteride (0.5mg); Drug: Harnal D Tablets and Harnal Capsules (both comprising 0.2 mg tamsulosin HCl)
- Dutasteride (0.5mg) (Experimental): Commercial formulation of dutasteride
  Interventions: Drug: FDC product of dutasteride (0.5mg) and tamsulosin HCl (0.2mg)
- Harnal-D Tablets and Harnal capsules (Experimental): Commercial formulations of Harnal-D Tablets and Harnal Capsules both comprising 0.2mg tamsulosin HCl
  Interventions: Drug: FDC product of dutasteride (0.5mg) and tamsulosin HCl (0.2mg)

INTERVENTIONS:
Drug: Dutasteride (0.5mg) — This study is an open-label, randomized, single dose, four-period cross-over study.
  Arms: Fixed dose combination product
Drug: FDC product of dutasteride (0.5mg) and tamsulosin HCl (0.2mg) — FDC (with 10% enteric coated tamsulosin pellets); (2): FDC (with 15% enteric coated tamsulosin pellets);
  Arms: Dutasteride (0.5mg); Harnal-D Tablets and Harnal capsules
Drug: Harnal D Tablets and Harnal Capsules (both comprising 0.2 mg tamsulosin HCl) — a commercial formulation of dutasteride plus tamsulosin HCl (Harnal-D Tablet); (4): a commercial formulation of dutasteride plus tamsulosin HCl(Harnal Capsule). Each dosing session will be separated by a wash-out period of 5 to 10 days
  Arms: Fixed dose combination product

SUMMARY:
This study aims to determine the relative bioavailability of tamsulosin hydrochloride in a fixed dose combination capsule of dutasteride and tamsulosin hydrochloride (0.5 mg/0.2 mg) relative to co-administration of dutasteride 0.5 mg capsules and tamsulosin hydrochloride 0.2 mg tablets or capsules. Two fixed dose combination capsules will be tested; one will contain tamsulosin hydrochloride pellets with a 15% enteric coating, and the other tamsulosin hydrochloride pellets with a 10% enteric coat. In addition, two formulations of tamsulosin hydrochloride will be tested in the co-administration with dutasteride 0.5 mg; a 0.2 mg oral disintegrating tablet and a 0.2 mg hard shell capsule. This will be an open-label, randomized, single dose, four-period crossover in healthy male subjects of North East Asian ancestry. Subjects will receive single oral doses in four treatment periods, each separated by a 5-10 day washout period. Blood samples for pharmacokinetic analysis will be taken at regular intervals after dosing. Safety will be assessed by measurement of blood pressure, heart rate and review of adverse events. The study will enrol approximately 30 healthy male subjects to ensure that 24 complete the study.

DETAILED DESCRIPTION:
This study is an open-label, randomized, single dose, four-period crossover study which aims to determine the relative bioavailability of tamsulosin hydrochloride in a fixed dose combination capsule of dutasteride and tamsulosin hydrochloride (0.5 mg/0.2 mg) relative to co-administration of dutasteride 0.5 mg capsules and tamsulosin hydrochloride 0.2 mg tablets or capsules. Two fixed dose combination capsules will be tested; one will contain tamsulosin hydrochloride pellets with a 15% enteric coating, and the other tamsulosin hydrochloride pellets with a 10% enteric coat. In addition, two formulations of tamsulosin hydrochloride will be tested in the co-administration with dutasteride 0.5 mg; a 0.2 mg oral disintegrating tablet and a 0.2 mg hard shell capsule. Subjects will receive single oral doses in four treatment periods, each separated by a 5-10 day washout period. Blood samples for pharmacokinetic analysis will be taken at regular intervals after dosing. Safety will be assessed by measurement of blood pressure, heart rate and review of adverse events. The study will enrol approximately 30 healthy male subjects to ensure that 24 complete the study.

BACKGROUND:

Dutasteride (AVODART ™) is an approved potent 5-alpha-reductase inhibitor indicated for the treatment of symptomatic benign prostatic hyperplasia (BPH) in men with an enlarged prostate to improve symptoms, reduce the risk of acute urinary retention and reduce the risk of the need for BPH-related surgery [AVODART Package Insert, 2009].

In humans, dutasteride is well-tolerated in single doses up to 40mg/day, multiple doses up to 40mg/day administered for 7 days, and 5 mg/day administered for 24 weeks. In single dose clinical studies, the overall incidence and type of adverse events (AEs) was similar across the dutasteride, placebo, and finasteride treatment groups.

Tamsulosin (Harnal, Harnal D, Flomax) is an alpha-1-adrenoceptor blocking agent approved for the treatment of signs and symptoms of benign prostatic hyperplasia. Tamsulosin HCl is extensively metabolized, with less than 10% of the dose excreted in the urine unchanged [Harnal, 2009; Harnal, 2011; Flomax, 2011]. In human liver microsomes and human lymphoblastoid cells expressing CYP cDNAs in vitro, tamsulosin HCl is metabolized by both CYP3A4 and CYP2D6 [Matsushima, 1998].

Clinical data exist to support that tamsulosin (an alpha-1-adrenoceptor antagonist), when used in combination with dutasteride (a 5-alpha reductase inhibitor), offers a more effective treatment for the symptoms of benign prostatic hyperplasia than either drug used alone [GSK study ARI40005, GlaxoSmithKline document number HM2002/00171/01]. In addition, data from a large, multi-centre National Institutes of Health-sponsored Medical Therapy of Prostatic Symptoms (MTOPS) study revealed greater benefits of combination alpha-1-adreoceptor antagonist and 5-alpha-reductase inhibitor therapy compared with either monotherapy in males with BPH [McConnell, 2002].

Clinical drug interaction studies have shown no pharmacokinetic or pharmacodynamic interactions between dutasteride and tamsulosin. Dutasteride may be administered with or without food. Tamsulosin should be administered with food. Food effect PK data exists for co-administration of dutasteride and tamsulosin given in a fixed dose combination (FDC) capsule formulation relative to the co-administration of the two components, dutasteride and tamsulosin HCl; GSK studies ARI109882, [GlaxoSmithKline document number ZM2007/00022/00], and ARI114694, [GlaxoSmithKline document number ZM2010/00028/00]. In the latter study, the dose of tamsulosin HCl administered was 0.2 mg versus 0.4mg administered in ARI109882. The dose of dutasteride was the same in both studies (0.5mg). In ARI109882, the GSK combination capsule was found to be bioequivalent (under both fed and fasted conditions) to the marketed products administered separately. ARI114694 demonstrated bioequivalence for dutasteride but not for tamsulosin when administered as an FDC product (of dutasteride 0.5 mg and tamsulosin 0.2 mg) relative to co-administration of separate commercial formulations of dutasteride (0.5 mg) and tamsulosin (0.2 mg) in the fed and fasted stage in different North East Asian ethnic groups.

This study aims to investigate the bioequivalence of tamsulosin only by investigating two different FDC formulations with 10 % or 15% Enteric Coated Tamsulosin pellets (0.2 mg) and Dutasteride 0.5 mg relative to co-administration of a commercial formulation of dutasteride (0.5 mg) and two different commercial formulations of 0.2 mg tamsulosin,Harnal Capsule and Harnal-D Tablet. Specifically, the study aims to investigate the bioavailability of the following:

* FDC (with 10% enteric coated tamsulosin pellets) to a commercial formulation of dutasteride plus tamsulosin (Harnal-D Tablet)
* FDC (with 10% enteric coated tamsulosin pellets) to a commercial formulation of dutasteride plus tamsulosin (Harnal Capsule)
* FDC (with 15% enteric coated tamsulosin pellets) to a commercial formulation of dutasteride plus tamsulosin (Harnal-D Tablet) (also investigated in ARI114694)
* FDC (with 15% enteric coated tamsulosin pellets) to a commercial formulation of dutasteride plus tamsulosin (Harnal Capsule) Both Harnal-D tablets and Harnal capsules are included as comparators as bioequivalence of the 10 or 15 % FDC formulations to Harnal Capsules would provide a registration pathway for China, where Harnal Capsules are commercially available. As Harnal capsules are not available in Korea and Japan, bioequivalence to Harnal-D tablets would allow the FDC to be registered in China, Korea and Japan, where Harnal-D tablets are approved.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Males between 20 and 45 years of age inclusive, at the time of signing the informed consent form.
* Japanese ancestry defined as being born in Japan, having four ethnic Japanese grandparents, holding a Japanese passport or identity papers and being able to speak Japanese, or Korean ancestry defined as being born in Korea, having four ethnic Korean grandparents, holding a Korean passport or identity papers and being able to speak Korean, or Chinese ancestry defined as being born in China, Hong Kong, Singapore or Taiwan, having four ethnic Chinese grandparents, holding a Chinese passport or identity papers and being able to speak Chinese.

Japanese, Korean and Chinese subjects should also have lived outside their respective countries for less than 10 years.

* Male subjects with female partners of child-bearing potential must agree to use one of the protocol-approved contraception methods .This must be followed from the time of the first dose of study medication until 45 days after the last dose.
* BMI within the range 18 -28 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Single QTcB < 450 msec
* AST, ALT, alkaline phosphatase and bilirubin less than or equal to 1.5xULN (isolated bilirubin greater than 1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin is less than 35%).

Exclusion Criteria:

Medical Condition Exclusions:

* Poor metabolizer for CYP2D6 substrates as determined by genotyping of selected CYP2D6 variants at screening.
* History of postural hypotension, dizziness, poor hydration, vertigo, vaso-vagal reactions or any other signs and symptoms of orthostasis, which in the opinion of the investigator could be exacerbated by tamsulosin and result in putting the subject at risk of injury.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* A positive test for HIV antibody.
* Subject is mentally or legally incapacitated.

Medical Exclusions:

* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort, Black Khosh, Dong Quai, Milk Thistle, licorice) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to tamsulosin hydrochloride or durasteride, components thereof or drugs of this class or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* A history of sensitivity to heparin or heparin-induced thrombocytopenia
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Lifestyle Exclusions:

* A positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* History of regular alcohol consumption within 6 months of the screening visit defined by the following Australian guidelines:

Males: An average weekly intake greater than 21 units or an average daily intake greater than 3 units. One unit is equivalent to 270 mL of full strength beer, 470 mL of light beer, 30 mL of spirits and 100 mL of wine.

Subjects must be able and willing to abstain from beverages and foods containing alcohol 24 hours prior to and during the dosing day.

* Consumption of red wine, grapefruit juice, grapefruit and related hybrids from 7 days prior to the first dose of study medication.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2011-06-30 (Actual); Primary Completion 2011-09-07 (Actual); Study Completion 2011-09-07 (Actual)

PRIMARY OUTCOMES:
Bioavailability of tamsulosin in 2 FDC formulations (Tamsulosin 0.2 mg and Dutasteride 0.5 mg) relative to co-administration of AVODART capsules with Harnal-D tablets or Harnal capsules in male subjects of Asian ancestry in the fed state | From dosing to 72 hours post-dose

SECONDARY OUTCOMES:
Bioavailability of tamsulosin in one FDC formulation relative to the other FDC formulation (each capsule containing 0.2 mg tamsulosin HCl and 0.5 mg dutasteride) in healthy male subjects of Asian ancestry in the fed state. | From dosing to 72 hours post-dose
Safety and tolerability of dosing with one FDC formulation relative to the other FDC formulation (each capsule containing 0.2 mg tamsulosin HCl and 0.5 mg dutasteride) in healthy male subjects of Asian ancestry in the fed state | Vital signs from dosing to 72 hr post-dose. Adverse events monitoring from dosing to 72hr post-dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] AVODART (Dutasteride 0.5 mg) Product Information. February, 2009.
- [Background] FLOMAX (Tamsulosin hydrochloride) Product Information. January, 2011.
- [Background] GlaxoSmithKline Document Number 2011N112801_00 Study ID ARI114694. GlaxoSmithKline studyARI114694: An open-label, randomized, single dose, two-period crossover study to determine the bioavailability of a fixed dose combination capsule formulation of dutasteride and tamsulosin hydrochloride (0.5 mg/0.2mg) relative to co-administration of dutasteride 0.5mg capsules and tamsulosin hydrochloride 0.2mg tablets in healthy male subjects of north east Asian and non-Asian ancestry;. Report Date 02-May-2011.
- [Background] GlaxoSmithKline Document Number HM2002/00171/01 Study ID ARI40005. A randomised, double-blind, parallel group study to investigate the efficacy and safety of treatment with Dutasteride (0.5mg) and Tamsulosin (0.4mg), administered once daily for 4 years, alone and in combination, on the improvement of symptoms and clinical outcome in men with moderate to severe symptomatic benign prostatic hyperplasia;. Report Date 09-Jul-2004.
- [Background] GlaxoSmithKline Document Number ZM2007/00022/00 Study ID ARI109882. An Open-Label, Randomized, Single Dose, Three-Period Crossover Study to Determine the Bioequivalence and Food Effect of a Combination Capsule Formulation of Dutasteride and Tamsulosin Hydrochloride (0.5mg/0.4mg) Compared to Concomitant Dosing of AVODART 0.5mg and FLOMAX 0.4 mg Commercial Capsules in Healthy Male Subjects. Report Date 30-Aug-2007.
- [Background] HARNAL (Tamsulosin hydrochloride 0.2 mg) Product Information. , 2011.
- [Background] HARNAL-D (Tamsulosin hydrochloride 0.2 mg) Product Information. , 2009.
- [Background] Matsushima H, Kamimura H, Soeishi Y, Watanabe T, Higuchi S, Tsunoo M. Pharmacokinetics and plasma protein binding of tamsulosin hydrochloride in rats, dogs, and humans. Drug Metab Dispos. 1998 Mar;26(3):240-5. PMID 9492387
- [Background] McConnell JD. The long term effects of medical therapy on the progression of BPH: Results from the MTOPS Trial (abstract 1042). 167 (4):265, 2002. J. Urology. 2002;167 (4):265.
- See also: Results for study 115707 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/115707?search=study&study_ids=115707#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 115707 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115707 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115707 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115707 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115707 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115707 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115707 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register